CLINICAL TRIAL: NCT02269371
Title: Auricular Acupuncture in the Treatment of Obesity: a Randomized, Placebo-controlled, Trial
Brief Title: Auricular Acupuncture in the Treatment of Obesity
Acronym: AcupObesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Crawford, Principal Investigator, Mike O'Callaghan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20140089H
Record Dates: First submitted 2014-10-14; First posted 2014-10-21 (Estimated); Results first posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Acupuncture, Ear; Acupuncture Therapy; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Group 1: Standard of care weight loss intervention plus auricular acupuncture at Shen Men, Point Zero, and Appetite Control Point/Hunger Point in each ear.
  Interventions: Other: Auricular Acupuncture
- Group 2 (Sham Comparator): Group 2: Standard of care weight loss intervention plus sham acupuncture at three nonacupoints in each ear.
  Interventions: Other: Sham Acupuncture

INTERVENTIONS:
Other: Auricular Acupuncture — Standard of care weight loss intervention plus auricular acupuncture at Shen Men, Point Zero, and Appetite Control Point/Hunger Point in each ear.
  Other Names: acupuncture
  Arms: Group 1
Other: Sham Acupuncture — Standard of care weight loss intervention plus sham acupuncture at three nonacupoints in each ear.
  Other Names: sham
  Arms: Group 2

SUMMARY:
Male and female DoD beneficiaries ages 18 years or older, who are referred for a standard of care weight loss intervention for treatment of obesity will be recruited. Subjects will be randomized into one of two groups receiving either a standard of care weight loss intervention plus auricular acupuncture at Shen Men, Point Zero, and Appetite Control Point/Hunger Point or receiving a standard of care weight loss intervention plus sham auricular acupuncture. Subjects will receive treatment in accordance with their randomization group for 12 weeks then have one additional follow up visit at week 24. The following measures will be obtained: height, weight, waist circumference, and Body Mass Index will be calculated.

DETAILED DESCRIPTION:
Screening Visit:

Obtain signed Informed Consent document and HIPAA Authorization. Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) to verify the inclusion/exclusion criteria and to verify the inclusion/exclusion criteria including previous encounter, vital signs review, medication list, co-morbidities, demographics, problems list, and note any prior acupuncture received.

Record: Date of birth, age, gender, race, ethnicity, last 4 of social security number, name of standard of care weight loss intervention, current email address, height (in inches), weight (in pounds), waist circumference (in inches) measurement, previous bariatric surgery, and body mass index calculated.

Visit 1-Week 1: (1st week of standard of care weight intervention)

Subjects will be randomized into 1 of 2 groups and treated:

* Group 1: Standard of care weight loss intervention plus auricular acupuncture at Shen Men, Point Zero, and Appetite Control Point/Hunger Point in each ear. The 3 needles will remain in each ear for 15 minutes.
* Group 2: Standard of care weight loss intervention plus sham acupuncture at three nonacupoints in each ear. The 3 needles will remain in each ear for 15 minutes.

All subjects, regardless of randomization group, will be instructed to have no heavy meals, no excessive hot or cold foods, no heavy exercise or intercourse, and no alcohol for 24 hours after this visit.

Visit 2-12 (Week 2-12 of standard of care weight intervention):

Subjects will be given treatment according to their randomization group. The acupuncture needles will be applied and remain in each ear for 15 minutes.

Record: weight, waist circumference measurement, and document compliance for standard of care weight loss intervention (i.e. attendance and measurements from class).

All subjects, regardless of randomization group, will be instructed to have no heavy meals, no excessive hot or cold foods, no heavy exercise or intercourse, and no alcohol for 24 hours after this visit.

Visit 13 (Week 24/12 weeks post visit 12):

Record: weight, and waist circumference measurement.

Subjects will be asked the following questions:

* Do you follow a regular routine of physical exercise? Yes/No *If yes, what type of exercise (mark all that apply):
* Aerobic (cardiovascular endurance, e.g. cycling, swimming, walking, hiking)
* Anaerobic (strength or resistance, e.g. weight lifting, sprinting, interval training)
* Flexibility (stretching, e.g. yoga, pilates, gymnastics) On average, how many times per week do you exercise?

  * 0-1
  * 2-4
  * 5+ How many minutes on average is each exercise session?
  * 10-20
  * 20-30
  * 30-60
  * 60 At what level of intensity?
  * Light
  * Moderate
  * Heavy How would you rate the "health" of your eating habits?
  * Poor
  * Fair
  * Average
  * Good
  * Excellent

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

Male and female DoD beneficiaries, aged 18 years or older, with a Body Mass Index of 30 or greater who were referred to a standard of care weight loss intervention

Exclusion:

Pregnant women Patients who are taking weight loss medication Uncontrolled hypothyroidism Absence of their ear Active cellulitis of their ear Ear anatomy precluding identification of acupuncture landmarks and use of hearing aids that preclude the insertion of needles

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinton Borchardt, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Hospital/Nellis Air Force Base, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Male and female Department of Defense beneficiaries ages 18 years or older were recruited at the Mike O'Callaghan Federal Medical Center. No special populations were recruited. The recruitment began April 2015 and ended February 2016.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 46 | 36
Completed | 29 | 25
Not Completed | 17 | 11

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (Auricular Acupuncture): Group 1: Standard of care weight loss intervention plus auricular acupuncture at Shen Men, Point Zero, and Appetite Control Point/Hunger Point in each ear.
  Auricular Acupuncture: Standard of care weight loss intervention plus auricular acupuncture at Shen Men, Point Zero, and Appetite Control Point/Hunger Point in each ear.
- Group 2 (Sham Acupuncture): Group 2: Standard of care weight loss intervention plus sham acupuncture at three nonacupoints in each ear.
  Sham Acupuncture: Standard of care weight loss intervention plus sham acupuncture at three nonacupoints in each ear.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Auricular Acupuncture) | Group 2 (Sham Acupuncture) | Total
Number analyzed (Participants) | 46 | 36 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 31 | 69
  >=65 years | 8 | 5 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 19 | 46
  Male | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Weight Change
Description: As assessed by weight in pounds. Weight change between baseline and week 24. Positive number equals pounds lost.
Time Frame: baseline to week 24 (12 wks post visit 12)
Population: participants analyzed are those who completed the study and did not withdraw
Measure: Mean (Full Range); unit: pounds
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 25 | 26
pounds | 7 [0 to 42.4] | 15.1 [0 to 37.4]

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/36
Other Adverse Events (participants affected / at risk) | 0/46 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes